CLINICAL TRIAL: NCT03212547
Title: The Effect of a Neonatologist's Standardized Guidance Intervention on Late and Moderately Late Preterm Infants With Sustained Social Withdrawal: a Randomized Controlled Trial in Chile.
Brief Title: The Effect of a Neonatologist's Standardized Guidance Intervention on Preterm Infants With Relational Withdrawal.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Clinica Alemana de Santiago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADBB Chile
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Social Withdrawal of Childhood or Adolescence; Preterm Infant
Keywords: ADBB; social withdrawal behavior; preterm; posttraumatic stress; postpartum depression; early detection; interactional guidance; synchronization within parent infant interaction
MeSH Terms: conditions — Premature Birth; Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants: The families of the MLP infants will remain blind to the group they belong to. Families will receive feedback on their infant's ADBB scores only after the final assessment (12 months).
  Care providers: neonatologists who care for participants during the trial are aware if the participants enter to the experimental or control group.
  Investigator: the principal investigator (JB) is also an external evaluator. He is an ADBB- trained psychologist who doesn't participate in the follow-up of any of the participants. He is blind to the ADBB scores of the ADB- trained neonatologists.
  Outcome assessment: Regarding to the ADBB assessment, once the ADBB score is assigned, this data is collected by a study coordinator, also blind to the group category.
  Data collection assessors: They are not trained in the ADBB scale, and don't have contact with the participants or their families.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Verbal interventions made on infants (accompanied by their mothers) who presents sustained social withdrawal detected on the child consultations (at 2, 6 and 12 months of corrected gestational age), made by neonatologists certifieds in the assess of Alarm Distress Baby Scale. Theintervention is described in a guide for "Promotion of verbal interventions for interaction" , and will be supplemented with a written guideline for parents.
  Interventions: Behavioral: Verbal Intervention
- Control group (No Intervention): Control group: infants will assist at child consultations (at 2, 6 and 12 months of corrected gestational age) whit non trained neonatologists. However, these group will receive a development stimulation guide adapted of the ministerial guides for the stimulation of development of the Ministry of Health of Chile.

INTERVENTIONS:
Behavioral: Verbal Intervention — Promotion of verbal interventions:
  1. Detecting whether the infant has social withdrawal.
  2. The physician will verbally intervene.
  3. Positive response (+) from the infant, the evaluator will point out this to the parents.
  4. Negative response (-) from the infant, the evaluator will include the parents in the interaction.
  5. If he infant establishes positive contact (+) with the parents, he/she will point out this response to them.
  6. If the infant does not establish positive contact (-)with the parents, repeat step 2.
  7. If the infant offers a positive response (+) to the second attempt of verbal intervention, the evaluator will point out this response to the parents.
  8. At the end of each medical check-up, give and explain the "ADBB Intervention Sheet".
  Arms: Experimental group

SUMMARY:
The objective of this project is to determine the effect of the verbal intervention on the decrease in sustained social withdrawal in late and moderately late preterm infants. The intervention will be performed by pediatricians trained in the Alarm Distress Baby Scale (ADBB). This scale has been applied to term and preterm newborns in multiple international studies, but it has not yet been applied in Chile, nor with moderately late and late preterm infants.

Infants are social beings who are born with innate reciprocal communication skills that can be observed during the two first months after delivery in babies with normal development. These skills include abilities to make and maintain eye contact, to vocalize and to use facial expressions, body and head movements to start interactions. Micro-analytical studies have demonstrated the frequent appearance of short episodes of social withdrawal affecting the infant during mother-baby interactions, whose function is to regulate the interaction flow. This behavior can be perceived when the infant needs to calm down or when is tired, and as a reaction to transitory interaction disturbances. In contrast with these short episodes of social withdrawal, the occurrence of sustained social withdrawal in infants is significantly less and is frequently associated with pathological conditions, such as autism spectrum disorder, child depression, and severe or chronic pain. Additionally, sustained social withdrawal is a symptom of anxiety and post-traumatic stress disorders. Different studies have revealed a prevalence of 11-22% in pre-term infant populations. In addition, the increase in sustained social withdrawal has been related to deviations of the interaction skills, attachment, as well as to relational and behavioral disorders. The increase and chronification of sustained social withdrawal, used as a defensive conduct, imply a risk to the adequate development of an infant's potential and raise the probability of alterations in the development of his psychopathology.

DETAILED DESCRIPTION:
Patients and methods: a prospective multicenter (Clínica Alemana de Santiago and Hospital San José) cohort randomized controlled trial. The study will comprise four periods (during hospitalization and at 2, 6 and 12 months of corrected age). An experimental and a control group will be randomized during the MLP newborn neonatal care unit hospitalization. The experimental group will be composed of late and moderately late preterm infants (MLP) born between 32 to 366 weeks of pregnancy, who will be verbally intervened by neonatologists in outpatient well child consultations at 2, 6 and 12 months corrected age, trough a standarized guidance intervention with the aim of potentiating the interaction of the infant with the parents to reduce sustained social withdrawal. Likewise, an analysis of both institutions (Clinica Alemana de Santiago and Hospital San Jose) will be performed to assess the differences between them. The tools that will be applied are the ADBB scale, as dependent variable; the Edinburgh Post-natal Depression Scale to be applied to parents; the Modified Perinatal Post-Traumatic Stress Disorder Questionnaire and the Revised Impact of Events Scale. During the hospitalization of MLP infants, the painful and invasive procedures to which the infant is subjected will be quantified, as well as neonatal pain, hours of skin-to-skin contact, breastfeeding and parental visits. Results relevance and applicability: Efficient early detection and intervention in infants with sustained social withdrawal behavior is essential to prevent problems in their social and emotional development. Assessing sustained social withdrawal using a standardized and simple scale like the ADBB Scale will allow for monitoring the infant and implementing cost-effective interventions that will benefit him, his family and the society. Identifying the risk groups, i.e. with difficulties in the social and emotional development area, will allow us to optimize the follow-up and integral support programs according to the infants' health needs as well as to establish a care standard.

Intervention Experimental group: the intervention consist in verbal interventions on infants (accompanied by their mother/father) who presents sustained social withdrawal detected on the child consultations (at 2, 6 and 12 months of corrected gestational age). The sustained social withdrawal will be assessed by neonatologists certifieds in the assess of Alarm Distress Baby Scale (during the child consultation) and by certifieds external evaluator, by means of a video (8 to 12 minutes of extension) that will be recorder by the neonatologist and assessed by the external evaluator. If the trained neonatologist detect sustained social withdrawal he will perform the verbal intervention during the child consultation. If the neonatologist does not detect sustained social withdrawal during the pediatric check-up, but the certified external evaluator does when assessing the video, the patient will be contacted and will receive treatment within the time limits described (+- 30 days). Also, the verbal intervention is described in a guide for "Promotion of verbal interventions for interaction" , and will be supplemented with a written guideline for parents to promote adequate interaction between parents and infant.

Control group: infants will assist at child consultations (at 2, 6 and 12 months of corrected gestational age) whit non trained neonatologists. These neonatologists will record a video that will be assessed by certifieds external evaluators. Infants in the control group won't receive the verbal intervention. However, they will receive a development stimulation guide adapted of the ministerial guides for the stimulation of development of the Ministry of Health of Chile.

Infants will be randomized while they are hospitalized in the NICU of Clinica Alemana de Santiago or in the NICU of Hospital San Jose. At the time of randomization, it will be defined whether the infant should attend medical check-ups at 2, 6 and 12 months of corrected gestational age with a neonatologists trained in Alarm Distress Baby Scale, or with a physician not trained, who will not perform the treatment.

Additionally, if during the experimental group medical check-ups at 2, 6 or 12 months of CGA, the physician trained in ADBB detects social withdrawal or finds any acute morbidity such as acute respiratory infection, fever, dehydration, hyperemesis, diarrhea, prolonged pain or irritability, or some acute condition that might affect the quality of the baby's interactions, he will perform a second assessment with the ADBB scale within 15 days.

At the end of the clinical trial, all the infants who present sustained social withdrawal in the medical check-up at 12 months of corrected gestational age will be offered free assessment and intervention (3 sessions) by the research team of this study.

ELIGIBILITY:
Inclusion Criteria:

* 32 to 36+6 week preterm chilean newborn. Gestational age assigned by neonatologist at birth.
* Spanish speaking parents.
* Parents with stable cohabiting and both of them responsible for the care of the infant
* Double or single pregnancy (monochorionic or bichorionic).
* Born and hospitalized within the first 48 hours of life or with a stay of at least 48 hours at Clínica Alemana de Santiago or at Hospital San José.
* Signed informed consent.

Exclusion Criteria:

* Mother with antecedents or confirmed exposure to cocaine, marihuana or cocaine crack during pregnancy
* Neurological disease that impairs the infant's development confirmed at birth.
* Major congenital malformations or genetic diseases suspected or confirmed antenatally or at birth.
* Perinatal asphyxia: <3 Apgar score at 1 minute or < 5 at 5 minutes and/or cord pH <7.0

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2017-09-19 (Actual); Primary Completion 2020-05-19 (Estimated); Study Completion 2020-07-19 (Estimated)

PRIMARY OUTCOMES:
Sustained social withdrawal | From date of the 2 months of corrected age medical checkup untill the date of the 12 months of corrected age medical checkup
  Quantitative categorical variable, ordinal. Category according sum of obtained scores (0-4: No withdrawal, 5-9: moderate withdrawal, 10 or more: Severe withdrawal).

SECONDARY OUTCOMES:
Post-partum depression | From date of the 2 months of corrected age medical checkup untill the date of the 12 months of corrected age medical checkup
  Quantitative categorical variable, nominal. Category obtained from scores lower or higher than 12 points in Edinburgh scale ("No risk" and "risk").
Post-traumatic stress symptoms | From date of the 2 months of corrected age medical checkup untill the date of the 12 months of corrected age medical checkup
  Quantitative categorical variable, nominal. Category obtained from scores lower or higher than 19 points in Modified Perinatal Post-traumatic Stress Disorder Questionnaire ("no risk" and "risk").
  Category obtained from scores lower or higher than 24 ("clinical concern") in Impact of Event Scale Revised (IES-R).
Premature infant pain | From date of admission to the NICU untill the date of medical discharge from the NICU or date of death from any cause, whichever came first, assessed up to 10 months
  Quantitative categorical variable, nominal. Categorys obtained from scores between 0 and 5 points (no pain), 6 and 11 points (pain) and 12 or more points (moderate to severe pain) in the "Premature Infant Pain Profile (PIPP)".
Painful invasive procedures | From date of admission to the NICU untill the date of medical discharge from the NICU or date of death from any cause, whichever came first, assessed up to 10 months
  Quantitative variable. Sum of the daily number of painful invasive procedures registered on the medical chart
Parental visiting time | From date of admission to the NICU untill the date of medical discharge from the NICU or date of death from any cause, whichever came first, assessed up to 10 months
  Quantitative variable. Sum of the daily minutes that the parents are visiting their preterm infants on the NICU
Breastfeeding time | From date of admission to the NICU untill the date of medical discharge from the NICU or date of death from any cause, whichever came first, assessed up to 10 months
  Quantitative variable. Sum of the daily minutes that the mothers are breastfeeding their preterm infants on the NICU
Skin to skin contact time | From date of admission to the NICU untill the date of medical discharge from the NICU or date of death from any cause, whichever came first, assessed up to 10 months
  Quantitative variable. Sum of the daily minutes that the parents are in skin to skin contact with their preterm infants on the NICU

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Bustamante Loyola, Phd student, Principal Investigator — Clínica Alemana de Santiago
Locations (1):
- Clinica Alemana de Santiago, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bustamante Loyola J, Perez Retamal M, Mendiburo-Seguel A, Guedeney AC, Salinas Gonzalez R, Munoz L, Cox Melane H, Gonzalez Mas JM, Simo Teufel S, Morgues Nudman M. The Impact of an Interactive Guidance Intervention on Sustained Social Withdrawal in Preterm Infants in Chile: Randomized Controlled Trial. Front Pediatr. 2022 Apr 1;10:803932. doi: 10.3389/fped.2022.803932. eCollection 2022. PMID 35433551
- [Derived] Bustamante Loyola J, Perez Retamal M, Morgues Nudman MI, Maturana A, Salinas Gonzalez R, Cox H, Gonzalez Mas JM, Munoz L, Lopez L, Mendiburo-Seguel A, Simo S, Palau Subiela P, Guedeney A. Interactive Guidance Intervention to Address Sustained Social Withdrawal in Preterm Infants in Chile: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Jun 26;9(6):e17943. doi: 10.2196/17943. PMID 32589156